CLINICAL TRIAL: NCT03545009
Title: Determination of the Independent Effects of Beetroot Juice Components, Dietary Nitrate and Antioxidants, on Exercise Tolerance and Health Benefits in Individuals With Obesity
Acronym: BEETIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gordon Fisher, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 300001210
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Disease; Obesity; Exercise
MeSH Terms: conditions — Metabolic Diseases; Obesity; Motor Activity | interventions — sodium nitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beetroot Juice (Experimental)
  Interventions: Dietary Supplement: Beetroot Juice
- Beetroot Juice no Nitrate (Active Comparator)
  Interventions: Dietary Supplement: Beetroot Juice no Nitrate
- Sodium Nitrate (Active Comparator)
  Interventions: Dietary Supplement: Sodium Nitrate
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Sodium Nitrate — 70ml sodium nitrate, matched for nitrate concentration in Beetroot Juice arm
  Arms: Sodium Nitrate
Dietary Supplement: Beetroot Juice no Nitrate — 70ml Concentrated Beetroot Juice with nitrate removed
  Arms: Beetroot Juice no Nitrate
Dietary Supplement: Beetroot Juice — 70ml Concentrated Beetroot Juice
  Arms: Beetroot Juice

SUMMARY:
The purpose of this study is to assess the effects of acute beetroot juice supplementation on exercise performance and cardiometabolic health in obese individuals with secondary cardiometabolic complications. Additionally, we will determine if the ergogenic health benefits of beetroot juice is due to the nitric oxide compound within the product, the antioxidant compound within the product, or a combination of the two compounds.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2
* Able to perform exercise testing on a cycle ergometer

Exclusion Criteria:

* Currently taking medications know to affect cardiovascular or respiratory function
* Currently supplementing with an antioxidant compound
* Current smoker
* Currently taking antibiotics
* Not willing to abstain from mouthwash use
* Currently participating in regular physical activity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Time to Exhaustion | A Time to Exhaustion Test will be conducted on each participant a total of four times throughout their participation in the study. This will take place approximately 2.5 hours post ingestion of the dietary supplement they are randomized to at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Fisher, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No